CLINICAL TRIAL: NCT01418521
Title: Safety and Effectiveness of a Balanced 3rd Generation HES Solution (Tetraspan®) Versus Albumin Solution for Volume Replacement in Patients After Cardiac Surgery
Brief Title: Safety and Effectiveness of a Balanced 3rd Generation HES Solution (Tetraspan®) After Cardiac Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Zvi Adler, Rambam Health Care Campus, cardiac surgery department
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RMB-0058.CTIL
Record Dates: First submitted 2011-08-09; First posted 2011-08-17 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2011-08

CONDITIONS: Elective Cardiac Surgery
Keywords: Cardiac surgery; Balanced 3rd generation Hydroxyethyl starch; Tetraspan; Ringer-albumin
MeSH Terms: interventions — Serum Albumin, Human

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ringer-albumin (Active Comparator): Patients receiving the standard care of ringer-albumin as volume replacement after cardiac surgery
  Interventions: Drug: Ringer- albumin
- Tetraspan (Experimental): patients receiving a 3rd generation HES solution (tetraspan) for volume replacement after cardiac surgery
  Interventions: Drug: Balanced hydroxyethyl starch solution

INTERVENTIONS:
Drug: Balanced hydroxyethyl starch solution — Patients receiving Tetraspan 6% ( a balanced 3rd generation Hydroxyethyl starch)for volume replacement after elective cardiac surgery as needed.
  Other Names: Tetraspan
  Arms: Tetraspan
Drug: Ringer- albumin — Patients receiving lactated ringer-albumin solution for volume replacement after cardiac surgery
  Other Names: HARTMANN Solution; Human albumin 20%- Zenalb
  Arms: Ringer-albumin

SUMMARY:
The purpose of this randomized controlled trial in patients undergoing cardiac surgery is to show that a 3rd generation HES (Hydroxyethyl Starch) solution - Tetraspan® is as good as in terms of safety and effectiveness as the commonly used albumin based solution for volume replacement after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained from the subject or his/her legal guardian before any assessment is performed.
* Male or Female subject, 18 years or older.
* Any elective cardiac surgery

Exclusion Criteria:

* Subjects with impaired liver function defined as an elevated level of ALT and AST over 100 U/L.
* Hyperhydration states (e.g. pulmonary edema, congestive heart failure).
* Renal failure with creatinine blood levels > 2.5 mg/dL or eGFR < 30 ml/min (calculated using the DMRD formula).
* Oliguria (UO<0.5ml\kg\hr) or anuria (not related to hypovolemia) more than 12 hours.
* Current Intracranial hemorrhage.
* Current, hard to balance hyperkalemia.
* Severe hypernatremia or severe hyperchloremia.
* Known hypersensitivity to hydroxyethyl starch or to any of the excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-08; Primary Completion 2013-07 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Chest tube drainage volume | Total volume at the time of removal of drains (48 hours after surgery on average)

SECONDARY OUTCOMES:
Volume of replacement fluids given after surgery at each group | Summary of volume replacement at the time of discharge from ICU (48 hours after surgery on average)
In hospital - all cause mortality | End of hospitalization (5 days postsurgery on average)
30-days all cause mortality | 30 days from surgery
Incidence of kidney injury as defined by RIFLE criteria | Duration of hospitalization after surgery (expected average duration of 5 days)
Incidence of coagulopathy as defined by prolonged PT\PTT and abnormal thromboelastogram not due to clotting inhibitors during hospitalization. | Duration of hospitalization after surgery (expected average duration of 5 days)
Volume of Transfused blood products during hospitalization postsurgery | Duration of hospitalization after surgery (expected average duration of 5 days)

CONTACTS AND LOCATIONS:
Overall Officials: Zvi Adler, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam health care campus, Haifa, Israel